CLINICAL TRIAL: NCT05476887
Title: An Open-label, Phase 2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of KP104 in Complement Inhibitor-naïve Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of KP104
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kira Pharmacenticals (US), LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KP104-201
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: KP104; Paroxysmal nocturnal hemoglobinuria; Complement Inhibitor; Dose Selection; Proof of Concept
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1: Dose escalation Cohort 1 (Experimental): Participants will receive escalating and varying dose intervals of KP104 every week.
  Interventions: Drug: KP104
- Part 1: Dose escalation Cohort 2 (Experimental): Participants will receive escalating and varying dose intervals of KP104 weekly or biweekly.
  Interventions: Drug: KP104
- Part 1: Dose escalation Cohort 3 (Experimental): Participants will receive escalating and varying dose intervals of KP104 weekly or biweekly.
  Interventions: Drug: KP104
- Part 2: Proof-of-concept Cohort 1 (Experimental): Participants will receive escalating and varying dose intervals of KP104 weekly or biweekly.
  Interventions: Drug: KP104
- Open-label extension (OLE) (Experimental): Participants will receive KP104, who benefit from KP104 treatment in Part 1 and 2
  Interventions: Drug: KP104

INTERVENTIONS:
Drug: KP104 — KP104 intravenously (IV loading + subcutaneous [SC] maintenance every week [QW] or every 2 weeks [Q2W]) will be administered.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, immunogenicity, pharmacokinetics, pharmacodynamics, and efficacy of KP104 in complement inhibitor-naïve participants with PNH. The study will be conducted in 2 parts. Part 1 is a dose-selection study to assess escalating doses and varying dose intervals of KP104. Part 2 is a proof-of-concept (POC) study assessing the efficacy of the optimal intravenous (IV) loading dose followed by the optimal maintenance dose and regimen of KP104. Participants who complete the Initial Treatment Period and demonstrate benefit from KP104 will be eligible for a 9-month open-label extension (OLE) treatment period.

ELIGIBILITY:
Inclusion Criteria:

Initial Treatment Period:

* Documented diagnosis of PNH confirmed by flow cytometry evaluation of white blood cells and red blood cells, with granulocyte or monocyte clone size of >= 10 percent (%) within 6 months of the Screening visit.
* Presence of 1 or more PNH-related signs or symptoms within 3 months of initiation of Screening.
* LDH >= 2.0 × upper limit of normal (ULN) at screening.
* Hemoglobin <= 10.0 g/dL at screening.
* Females of childbearing potential and males must practice effective contraception from Screening until 28 days after the end of study (EOS) visit.
* Females of childbearing potential must have a negative pregnancy test at Screening and within 24 hours prior to dosing of study drug.

Extension Treatment Period (OLE):

* Complete the 12-week (weekly dosing) or 13-week (biweekly dosing) Initial Treatment Period per the protocol.
* Benefited from KP104 treatment and will continue benefiting from KP104 treatment per the investigator's judgement.
* Willing to participate in Extension Treatment Period, able to comply with this protocol and be available for the entire duration of the study.

Exclusion Criteria:

Initial Treatment Period:

* Any clinically significant poorly controlled underlying illness other than PNH per discretion of investigators.
* Treatment of any infection with IV (within 30 days of Screening) or oral (within 14 days of Screening) antibiotics, antivirals, or antifungals.
* History of meningococcal infection.
* History of untreated tuberculosis.
* History of splenectomy
* Positive serology for Hepatitis C Virus (HCV) ribonucleic acid (RNA) or human immunodeficiency virus (HIV) at Screening
* History of bone marrow or stem cell transplantation
* Absolute neutrophil count (ANC) <500 cells per microliter (cells/μL)
* Reticulocyte count< 100 x 10^3 cells/μL
* Platelet count< 30,000 cells/μL
* History of systemic autoimmune disease
* Estimated glomerular filtration rate (eGFR) <30 milliliters/minute/1.73 meter square (mL/min/1.73 m^2) calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

Extension Treatment Period (OLE):

* Women who are pregnant.
* Women of childbearing potential and men with sexual partners of childbearing potential who are not using adequate contraception and who are not willing to use adequate contraception.
* Any medical condition that, in the opinion of the investigator, may pose a safety risk to a participant in this study, or may interfere with study participation.

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with Dose-limiting toxicities (DLT) | Up to Week 4
  A DLT is defined as any adverse event considered by the investigator to be KP104-related with a severity greater than or equal to (>=) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade 3 which also represents a shift from baseline clinical status of > 1 NCI CTCAE grade. A hypersensitivity/administration reaction occurring with a severity of Grade 2 despite the use of pre-medications will also be designated as a DLT.
Part 2: Percentage of participants with >= 2 grams per deciliter (g/dL) increase in hemoglobin level from Baseline in the absence of transfusion for weekly dosing | Baseline and at Week 12
  Blood samples will be collected for the analysis of increase in hemoglobin levels in the absence of transfusion.
Part 2: Percentage of participants with >= 2 g/dL increase in hemoglobin level from Baseline in the absence of transfusion for biweekly dosing | Baseline and at Week 13
  Blood samples will be collected for the analysis of increase in hemoglobin levels in the absence of transfusion.
Open-label Extension (OLE): Number of participants reporting Treatment Emergent Adverse Events (TEAEs), treatment-emergent serious adverse events (TESAEs) and AEs of special interest (AESIs) | Up to 9 months

SECONDARY OUTCOMES:
Part 2: Change from Baseline in serum lactate dehydrogenase (LDH) levels for weekly dosing | Baseline and at Week 12
  Blood samples will be collected for the analysis of serum LDH.
Part 2: Change from Baseline in serum LDH levels for biweekly dosing | Baseline and at Week 13
  Blood samples will be collected for the analysis of serum LDH.
Part 2: Change from Baseline in hemoglobin level for weekly dosing | Baseline and at Week 12
  Blood samples will be collected for the analysis of hemoglobin level
Part 2: Change from Baseline in the hemoglobin level for biweekly dosing | Baseline and at Week 13
  Blood samples will be collected for the analysis of hemoglobin level.
Part 2: Change from Baseline in red blood cell (RBC) transfusion dependence for weekly dosing | Baseline and at Week 12
  The RBC transfusion dependence is the difference in the volume of RBC transfusions per month for the 3 months prior to initiation of investigational product versus the volume of RBC transfusions per month for each month on study.
Part 2: Change in RBC transfusion dependence for biweekly dosing | Baseline and at Week 13
  The RBC transfusion difference is the difference in the volume of RBC transfusions per month for the 3 months prior to initiation of investigational product versus the volume of RBC transfusions per month for each month on study.
Part 1 and 2: Number of participants reporting TEAEs, TESAEs and AESIs | Up to Week 13
Part 1 and 2: Concentration within one hour of end of infusion (CEOI) of KP104 | Up to Week 13
Part 1 and 2: Trough concentration (Ctrough) of KP104 | Up to Week 13

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing
  - Jiangsu Province Hospital, Nanjing
  - Chinese Academy of Medical Sciences Peking Union Medical College - Institute of Hematology Blood Diseases Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes